CLINICAL TRIAL: NCT00828477
Title: Evaluation of Comfort With the Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) Xibrom (Bromfenac Ophthalmic Solution) 0.09% and Nevanac (Nepafenac Ophthalmic Suspension) 0.1% Following Selective Laser Trabeculoplasty (SLT)
Brief Title: Evaluation of Comfort With Xibrom (Bromfenac Ophthalmic Solution)0.09% and Nevanac (Nepafenac Ophthalmic Suspension) 0.1% Following Selective Laser Trabeculoplasty (SLT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: Nate Kleinfeldt, Coburn-Kleinfeldt Eye Clinic
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0144
Record Dates: First submitted 2009-01-14; First posted 2009-01-26 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Intraocular Pressure
MeSH Terms: interventions — bromfenac; nepafenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Xibrom (bromfenac)
  Interventions: Drug: Xibrom
- 2 (Active Comparator): Nevanac (nepafenac)
  Interventions: Drug: Nevanac

INTERVENTIONS:
Drug: Xibrom — Xibrom: two times a day for seven days in the first eye.
  Other Names: bromfenac
  Arms: 1
Drug: Nevanac — Nevanac: three times a day for seven days in the second eye.
  Other Names: nepafenac
  Arms: 2

SUMMARY:
The objective of this study is to evaluate and compare the comfort of bromfenac or nepafenac following SLT.

DETAILED DESCRIPTION:
Open label, single armed, cross over controlled study to evaluate comfort and IOP (Intraocular Pressure) changes of specific NSAIDs post SLT. Patients (n= 25, total 50 eyes) scheduled to undergo bilateral Selective Laser Trabeculoplasty (SLT) will instill bromfenac in the first eye to undergo SLT, and the contra lateral eye will receive nepafenac.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old, either gender or any race.
* Diagnosis of open-angle glaucoma or ocular hypertension requiring laser trabeculoplasty.
* Completion of written and informed consent/authorization prior to any study related procedures.
* Able to follow study protocol and likely to complete study schedule.

Exclusion Criteria:

* Known sensitivity to NSAIDs.
* History of neovascular or ocular inflammatory disease.
* Current use of topical or systemic anti-inflammatory medications.
* Females of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Tolerability of study medication | 28 days

SECONDARY OUTCOMES:
Intraocular pressure changes | 28 days
Visual Acuity | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Nate Kleinfeldt, M.D, Principal Investigator — Coburn-Kleinfeldt Eye Clinic
Locations (1):
- Coburn-Kleinfeldt Eye Clinic, 3340 6 Mile Rd Livonia, Michigan, United States